CLINICAL TRIAL: NCT07164118
Title: Therapeutic Effects of Pranayama Breathing Technique and Deep Breathing Exercises on Pain and Anxiety After Abdominal Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Muaz Gulsen, dr lecturer, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CU-SBF-CB-07
Record Dates: First submitted 2025-08-28; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Abdominal Surgery
Keywords: abdominal surgery; deep breathing exercise; pranamaya; pain; anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: There are 3 groups: pranamaya group, deep breathing exercise group and control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Before the surgery, patients in the pranayama intervention group will be taught the Pranayama breathing technique.
  Individuals in the deep breathing exercise intervention group will be taught deep breathing exercises by the researcher before the surgical intervention.
  No application will be made to the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Patients will not be taught breathing exercises. Pain will be assessed with the VAS at the 6th, 12th, and 24th postoperative hours, and anxiety will be assessed with the STAI-II on the preoperative morning and before discharge.
- Pranayama Breathing Group (Experimental): Pranayama breathing techniques will be taught before surgery. Starting 4 hours after surgery, 8-10 minutes of breathing exercises will be repeated every 2 hours. Pain will be measured before and after the exercises and at 6, 12, and 24 hours postoperatively. Anxiety will be measured with the STAI-II on the morning of the preoperative period and before discharge.
  Interventions: Behavioral: Pranayama Breathing Exercise
- Deep Breathing Group (Experimental): Deep breathing exercises will be taught before surgery. Six repetitions will be performed every two hours, starting four hours after surgery. Pain will be assessed with a VAS before and after the exercise and at 6, 12, and 24 hours. Anxiety will be measured with the STAI-II on the morning of the preoperative period and before discharge.
  Interventions: Behavioral: Deep Breathing Exercise

INTERVENTIONS:
Behavioral: Pranayama Breathing Exercise — Pranayama breathing technique consisting of 6 cycles, demonstrated by the researcher before the operation, supported by the brochure, and lasting 8-10 minutes every 2 hours from the 4th post-operative hour.
  Arms: Pranayama Breathing Group
Behavioral: Deep Breathing Exercise — Deep breathing exercise, demonstrated one-on-one before surgery and supported by a guide, applied 6 times every 2 hours from the 4th post-operative hour onwards.
  Arms: Deep Breathing Group

SUMMARY:
This study will be conducted to evaluate the therapeutic effects of pranayama breathing technique and deep breathing exercises on pain and anxiety after abdominal surgery.

DETAILED DESCRIPTION:
Abdominal surgeries often present with significant pain and the need for analgesia, and inadequate pain control can lead to delayed wound healing, cognitive impairment, stress, and anxiety. Surgical patients frequently experience anxiety and moderate to severe pain during the perioperative period. Non-pharmacological methods provide significant support to pharmacological treatments during this period. Pranayama and deep breathing exercises stand out as effective methods that promote relaxation and reduce pain perception and anxiety. While the literature supports the positive effects of these techniques, studies on their use after abdominal surgery are limited. This research aims to fill this gap and demonstrate the benefits of non-pharmacological approaches in postoperative care.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65,
* Having undergone elective abdominal surgery,
* Having no communication difficulties,
* Having no cognitive problems,
* Having no psychiatric illness,
* Having not previously practiced breathing exercises,
* Agreeing to participate in the study,
* Having an American Society of Anesthesiology (ASA) rating of I, II, or III will be included in the sample group.

Exclusion Criteria:

* Patients who developed complications such as bleeding, anastomotic leakage, atelectasis, deep vein thrombosis, or pulmonary embolism in the postoperative period; who wished to withdraw from the study at any stage; or who required intensive care in the postoperative period will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Spielberger State-Trait Anxiety Inventory: | 5 months
  Spielberger State-Trait Anxiety Inventory: First developed by Spielberger and his colleagues in 1970, it was adapted into Turkish by Öner and Le Compte (1982), and its validity and reliability studies were conducted. This inventory consists of two subsections, each containing 20 items: State Anxiety (STAI-I) and Trait Anxiety (STAI-II). In the state anxiety section, participants select one of the following options: "not at all," "a little," "a lot," or "completely." In the trait anxiety section, participants respond with the following options: "almost never," "sometimes," "most of the time." The total score on the scale ranges from 20 to 80; higher scores indicate higher anxiety levels. In the study conducted by Günaydın and Oflaz (1998), anxiety scores were classified according to their levels and defined as 20-39 as "mild", 40-59 as "moderate", 60-79 as "high" and over 80 points as "panic level anxiety".
Visual Analog Scale (VAS) | 5 months
  Visual Analog Scale (VAS) The Visual Analog Scale (VAS) was designed in 1983 by Price and colleagues to assess pain intensity. This measurement tool consists of a 10-cm-long straight line with the words "no pain" at one end and "unbearable pain" at the other. The patient is asked to mark a point on the line corresponding to the intensity of the pain they are experiencing; this point is scored in centimeters from the beginning. The score is categorized as no pain for 0, mild for 1-4, moderate for 5-6, severe for 7-8, and extreme pain for 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Afsin State Hospital, Kahramanmaraş, Afşin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No